CLINICAL TRIAL: NCT04725032
Title: Comparison of the Effects of Total Intravenous Anesthesia and Balanced General Anesthesia on Flash Visual Evoked Potential Monitoring During Sellar Tumors Resection
Brief Title: Effects of Intravenous Anesthesia and Balanced Anesthesia on Flash Visual Evoked Potentials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: HX-A-023(2020)
Record Dates: First submitted 2021-01-14; First posted 2021-01-26 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Brain Tumor Adult
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sevoflurane-propofol balanced anesthesia (Experimental)
  Interventions: Drug: Sevoflurane
- propofol-based total intravenous anesthesia (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol will be administered for anesthesia maintenance in patients randomized to the propofol-based TIVA arm of the study. In order to record the VEPs, standard spiral electrodes or subcutaneous electrodes will be inserted subcutaneously around the visual area and the Nicolet Viking IV System will be used to monitor VEP during surgery.
  Arms: propofol-based total intravenous anesthesia
Drug: Sevoflurane — Balanced general anesthesia with sevoflurane will be administered for anesthesia maintenance in patients randomized to the balanced general anesthesia arm of the study. In order to record the VEPs, standard spiral electrodes or subcutaneous electrodes will be inserted subcutaneously around the visual area and the Nicolet Viking IV System will be used to monitor VEP during surgery.
  Arms: sevoflurane-propofol balanced anesthesia

SUMMARY:
Intraoperative flash visual evoked potentials (FVEPs) could monitor visual function during neurosurgery. There are fewer reports comparing the effects of sevoflurane-propofol balanced anesthesia and propofol-based total intravenous anesthesia under comparable bispectral index (BIS) levels on the amplitude and latency of flash visual evoked potentials (FVEPs) for sellar or parasellar tumors resection neurosurgeries.

DETAILED DESCRIPTION:
The overall incidence rate of sellar tumors is 10-20% of brain tumors. Most of the initial symptoms of this tumor are visual or visual impairment. One of the primary complications of these operations is visual impairment, which directly relates to the quality of patients' life. Flash visual evoked potentials (FVEPs) is an important means of intraoperative visual function evaluation under general anesthesia. Intraoperative visual function damage can be avoided or reduced by observing the changing of FVEPs waves to guide the choice of surgical path.

However, since the diversity of anesthetic drugs and methods, there is still a great uncertainty impact on FVEPs, which will interfere with the interpretation and judgment of surgeons and neuroelectrophysiological physicians respect to the changes of FVEPs amplitude and latency, and further affect the operation decision-making. Therefore, it is urgent to establish a perfect anesthesia method for intraoperative monitoring of FVEPs. Although total intravenous anesthesia has been widely accepted for FVEPs monitoring, there are still some limitations, such as the possibility of intraoperative body movement and cough due to the restriction of muscle relaxant use under electrophysiological monitoring, as well as the depression on FVEPs of high maintained dosage under total intravenous anesthesia. The purpose of this study was to investigate the feasibility of FVEPs monitoring during endoscopic sellar tumor resection under combined intravenous anesthesia compared with total intravenous anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years;
2. ASA I-III;
3. Elective sellar or parasellar tumors resection;
4. Informed written consent

Exclusion Criteria:

1. Preoperative visual acuity<0.3;
2. BMI>30kg/cm2;
3. Uncontrolled hypertension, diabetes or cardiac diseases;
4. Preoperative cognitive disorders;
5. Sedatives, alcohol or analgesic addiction history;
6. Allergy to drugs of this study or contact allergy to Silicone products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
N2 amplitudes of FVEPs | 90min after anesthesia induction
  N145-P100 of FVEPs wave

SECONDARY OUTCOMES:
P100 latencies of FVEPs | 30, 60 and 90min after anesthesia induction
  P100 latencies of FVEPs wave
The visual acuity | The day before surgery, and one day after operation.
  The visual acuity before and after operation.
The visual field | The day before surgery, and one day after operation.
  The field of patients before and after operation.
N2 amplitudes of FVEPs | 30 and 60 after anesthesia induction
  N145-P100 of FVEPs wave

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, M.D., Ph. D, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Enrolled subjects will be assigned a subject identification number